CLINICAL TRIAL: NCT07149441
Title: Efficacy and Mechanism of Fecal Microbiota Transplantation in the Treatment of Inflammatory Bowel Disease: an Open-label Randomized Controlled Study
Brief Title: Efficacy and Mechanism of FMT in the Treatment of Inflammatory Bowel Disease: an Open-label Randomized Controlled Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Chen QiYi, Director of department, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT-IBD
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Disease (Crohn&Amp;#39;s Disease and Ulcerative Colitis); Fecal Microbiota Transplantation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation; Infliximab; Biological Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biological agent +FMT (Experimental): 47 patients were treated with biological agents combined with fecal microbiota transplants (FMT). All patients were followed up for 52 weeks after discharge. To observe the curative effect of FMT capsule treatment on UC or CD symptom-related scores of subjects and its remodeling effect on intestinal flora and verify its safety.
  Interventions: Procedure: Fecal microbiota transplantation; Drug: infliximab
- Biological agent (Experimental): 47 patients were treated with biological agents. All patients were followed up for 52 weeks after discharge. To observe the curative effect of FMT capsule treatment on UC or CD symptom-related scores of subjects and its remodeling effect on intestinal flora and verify its safety.
  Interventions: Drug: infliximab

INTERVENTIONS:
Procedure: Fecal microbiota transplantation — Fecal microbiota transplantation (FMT) achieves the purpose of treating intestinal and extra-intestinal diseases by transplanting the functional microbes in the feces of healthy people into the patient's intestine through the upper or lower alimentary tract routes to rebuild the patient's intestinal microbiota.
  Arms: Biological agent +FMT
Drug: infliximab — Intravenous infusion of infliximab once every 8 weeks.
  Other Names: Biological agent

SUMMARY:
This study enrolled 94 patients with UC or CD. Two groups received either 8-week intestinal bacterial transplant capsule therapy or biological therapy, respectively. The control group received biological therapy alone, while the experimental group received biological therapy combined with FMT. Both groups were followed up for 52 weeks after discharge. The efficacy of FMT capsule therapy on the subjects' UC or CD symptom-related scores and its effect on remodeling the intestinal flora were observed, and its safety was verified.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis was UC or CD, and the diagnosis was based on clinical, endoscopic and pathological evidence.
* IBD should be diagnosed for at least 6 months to rule out the possibility of natural remission of new cases.
* Patients should be in mild to moderate active stage (UC: Mayo score 3-10; CD: CDAI score: 150-449)
* Biological agents (such as anti-TNF-α drugs, vedolizumab, etc.) were used in the past, but no clinical remission was achieved.
* Voluntary participation and signing of informed consent.
* Adults aged 18-65.
* Can tolerate oral enterobacteria transplantation capsule treatment.

Exclusion Criteria:

* The diagnosis was UC or CD, and the diagnosis was based on clinical, endoscopic and pathological evidence.
* IBD should be diagnosed for at least 6 months to rule out the possibility of natural remission of new cases.
* Patients should be in mild to moderate active stage (UC: Mayo score 3-10; CD: CDAI score: 150-449)
* Biological agents (such as anti-TNF-α drugs, vedolizumab, etc.) were used in the past, but no clinical remission was achieved.
* Voluntary participation and signing of informed consent.
* Adults aged 18-65.
* Can tolerate oral enterobacteria transplantation capsule treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Endoscopic remission rate | 14th and 52nd week after joining the group.
  UC is endoscopic Mayo score 0-1; CD is simple endoscopic score (SES-CD)<3 or no ulcer.
Clinical remission rate | 14th and 52nd week after joining the group.
  UC is defined as Mayo score ≤2, and no single score > 1; CD is defined as CDAI (Crohn's disease activity index) < 150.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No